CLINICAL TRIAL: NCT04996407
Title: Comparison Effect of Using Between Survival Thermal Blanket and Draping Fabric as Substitute for Perforated Blanket With Forced Air Warmer Usage as Perioperative Warmer : Study on Inadvertent Perioperative Hypotermia in Geratric Patients
Brief Title: Survival Thermal Blanket Versus Draping Fabric to Prevent Hypothermia in Geriatric Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IndonesiaUAnes108
Record Dates: First submitted 2021-07-13; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Hypothermia; Anesthesia
Keywords: perioperative hypothermia; geriatric; survival thermal blanket; draping fabric
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- survival thermal blanket (Active Comparator): Patient will be using survival thermal blanket as substitute for perforated blanket with forced air warmer during anesthesia
  Interventions: Device: survival thermal blanket; Device: draping fabric
- draping fabric (Active Comparator): Patient will be using draping fabrics as substitute for perforated blanket with forced air warmer during anesthesia
  Interventions: Device: survival thermal blanket; Device: draping fabric

INTERVENTIONS:
Device: survival thermal blanket — patients were given a thermal blanket
Device: draping fabric — Patients were given a draping fabric

SUMMARY:
This study compare effect of using survival thermal blanket and draping fabric as substitute for perforated blanket to reduce the incidence of inadvertent perioperative hypothermia in geriatric patients.

DETAILED DESCRIPTION:
Study design was randomized single blinded. Total of 126 geriatric subjects from March-April 2021 were allocated into survival thermal blanket group (n=63) dan draping fabric group (n=63). Preinduction temperature was measured using timpanic membrane termometer. Intraoperatively, temperature is measured using nasopharynx.Study design was randomized single blinded. Total of 126 geriatric subjects from March-April 2021 were allocated into survival thermal blanket group (n=63) dan draping fabric group (n=63). Preinduction temperature was measured using timpanic membrane termometer. Intraoperatively, temperature is measured using nasopharynx.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years old
* Physical status ASA 1-3
* Undergo elective surgery under general anesthesia with or without regional anesthesia

Exclusion Criteria:

* Thermoregulation disturbance
* Abnormal thyroid function
* Fever caused by infectious disease in 7 days prior to surgery
* Pre-induction hypothermia with temperature below 36 degree
* On routine antipiretic
* Unstable hemodynamic preoperative and intraoperative

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with hypothermia in survival thermal blanket group | Before induction
  Measure by nasopharyngeal thermometer
Number of participants with hypothermia in survival thermal blanket group | every 15 minute during anesthesia
  Measure by nasopharyngeal thermometer
Number of participants with hypothermia in survival thermal blanket group | end of surgery
  Measure by nasopharyngeal thermometer

SECONDARY OUTCOMES:
Number of participants with hypothermia in draping fabric group | Before induction
  Measure by nasopharyngeal thermometer
Number of participants with hypothermia in draping fabric group | every 15 minute during anesthesia
  Measure by nasopharyngeal thermometer
Number of participants with hypothermia in draping fabric group | end of surgery
  Measure by nasopharyngeal thermometer

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided